CLINICAL TRIAL: NCT03658486
Title: Exercise for Advanced Prostate Cancer: a Multicomponent Feasibility Trial in Men With Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Exercise for Advanced Prostate Cancer: a Multicomponent Feasibility Trial
Acronym: EXACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: HSC Public Health Agency (Unknown)
Responsible Party: Principal Investigator, Gillian Prue, Senior Lecturer, Queen's University, Belfast
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B18/15
Record Dates: First submitted 2018-08-16; First posted 2018-09-05 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer Metastatic; Castration-resistant Prostate Cancer
Keywords: Exercise; Metastatic castrate-resistant prostate cancer
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Other): 12 weeks of progressive, home-based, moderate intensity, aerobic and strengthening exercise. Aerobic exercise will be completed 5 days per week, commencing with a single 10 minute bout and progressing to 30 minutes of continuous brisk walking at week 12. Strengthening exercises will involve whole body activities and commence with 1 set of each exercise (8-15 repetitions) and progress to 3 sets. The strengthening exercises will gradually progress in difficulty throughout the program.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise programs will be individually tailored to the capabilities of each participant and gradually progressed accordingly. Each patient will be assigned a moderate intensity walking and strengthening program to complete at home. At baseline, 12 and 24 weeks patients will wear an accelerometer to determine activity levels. At these time points, patients will also complete a physical fitness assessment (timed sit-to-stand and six minute walking tests) and a range of quality of life questionnaires. At baseline, patients will receive a behaviour change consultation and continued support throughout the intervention. Each patient will receive a pedometer during the home-based, unsupervised regime to monitor step count and they are expected to complete a daily physical activity diary. Upon completion of the 24 week follow-up, patients will be invited to partake in semi-structured interviews to determine the effectiveness of the program and their experience throughout.

SUMMARY:
This feasibility study will investigate whether men with metastatic prostate cancer can take part in and progress through a home-based exercise program. This study will evaluate the effects of exercise on a range of disease and treatment-related outcomes.

DETAILED DESCRIPTION:
This 12 week multicomponent, tailored, progressive program will consist of both moderate intensity walking and strengthening exercises at home. This single centre, single arm study will incorporate a behavioural change consultation at baseline and weekly behavioural support throughout. This study will follow-up patients at 24 weeks to determine exercise maintenance. Outcome measures will be completed at baseline, 12 and 24 weeks. A qualitative evaluation will be conducted after the 24 week follow-up to determine impact, patient experience and measures that might assist in refining the program.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate with progressive systemic metastatic disease despite castrate levels of testosterone (<50ng/dL).
* At enrolment, patients must have demonstrated progressive disease since the most recent change in therapy.
* Patients must be on ADT with a GnRH agonist/antagonist or prior bilateral orchiectomy. All patients must be on ADT during the study period.
* ≥ 4 weeks since last surgery and fully recovered.
* No known contraindications to moderate intensity exercise such as (but not limited to) brain metastases, acute congestive heart failure, unstable angina, serious or non-healing wound, peripheral neuropathy greater than or equal to Grade 3. Recent myocardial infarction.
* Age ≥ 18 years.
* ECOG performance status 0-2.
* Medical clearance by treating clinician.

Exclusion Criteria:

* Men currently exceeding ACSM recommended exercise guidelines (150 mins of moderate and/or 60 mins of high intensity exercise per week).
* Men with brain metastases.
* Men with a currently active second malignancy other than non-melanoma skin cancer.
* Congestive heart failure or recent serious cardiovascular event.
* Chest pain brought on by physical activity.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility - recruitment. | At baseline.
  The number of participants that agree to participate or are excluded.
Feasibility - adherence to the exercise intervention. | Throughout the 24 week study period.
  Determine the percentage of patients adhering to the program and the weekly behavioral consultation sessions.
Feasibility - attrition rates. | Throughout the 24 week study period.
  The number of patients that withdraw.
Feasibility - safety / adverse events. | Monitored throughout the 24 week study period.
  Any safety / adverse events, in general or in relation to the exercise program, will be documented by the research team.
Feasibility - patient experience. | Following the study conclusion at 24 weeks.
  Determined by qualitative evaluation, using semi-structured interviews, to assess experiences, accessibility and acceptability of the exercise intervention.

SECONDARY OUTCOMES:
Anthropometric assessment. | At baseline, 12 and 24 weeks.
  Height will be measured in cm and body weight in kg, which will be combined to report BMI in kg/m(squared).
Hip and waist circumference analysis. | At baseline, 12 and 24 weeks.
  Hip and waist circumference will be measured in cms.
Functional ability assessment. | At baseline, 12 and 24 weeks.
  The amount of repetitions achieved during a 30 second sit-to-stand test will be recorded.
Physical fitness assessment. | At baseline, 12 and 24 weeks.
  Distance covered in meters during a six minute walk test will be recorded.
Objectively measure of physical activity levels. | At baseline, 12 and 24 weeks.
  Patients will wear an accelerometer for 7 full days.
Perceived physical activity levels. | At baseline, 12 and 24 weeks.
  Patients will complete an International Physical Activity Questionnaire (IPAQ-SF). This questionnaire will comprise 4 generic items to obtain comparable health-related physical activity. Patients will detail the number of days, hours and minutes that they undertake (1) vigorous exercise (2) moderate exercise (3) walking exercise and (4) sitting. Total physical activity will be generated and monitored for improvement or decline.
Cancer-related fatigue by questionnaire. | At baseline, 12 and 24 weeks.
  Fatigue will be measured by the Functional Assessment of Cancer Therapy - Fatigue (FACIT-Fatigue) questionnaire. Patients will score several fatigue items over the past 7 days on a scale (0 = not at all; 4 = very much), generating a total (0 - 52) with higher scores linked to greater quality of life.
Quality of life will be measured using a questionnaire. | At baseline, 12 and 24 weeks.
  Quality of life will be measured by the Functional Assessment of Cancer Therapy - Prostate (FACT-P) questionnaire. Patients will score a series of questions (0 = not at all; 4 = very much) in five sections (physical well-being; social/family well-being; emotional well-being; functional well-being; additional concerns) for the past 7 days. Higher scores will suggest better quality of life.
Quality of life will be measured using questionnaires. | At baseline, 12 and 24 weeks.
  Quality of life will be measured by the EuroQOL Five Dimension Questionnaire (EQ5D). Patients will select a level of difficulty (I have no - I have extreme) on that particular days health for mobility, self-care, usual activities, pain / discomfort and anxiety / depression. Patients will then rate 'how good' or 'how bad' their health is on that day using a 100 point scale (0 = worst health you can imagine; 100 = best health you can imagine).
Pain will be measured through a questionnaire. | At baseline, 12 and 24 weeks.
  Bone pain will be monitored using the Brief Pain Inventory Short Form (BPI-SF).

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Ireland Cancer Centre, Belfast City Hospital, Belfast, United Kingdom

REFERENCES:
- [Derived] Brown M, Murphy M, McDermott L, McAneney H, O'Sullivan JM, Jain S, Prue G. Exercise for advanced prostate cancer: a multicomponent, feasibility, trial protocol for men with metastatic castrate-resistant prostate cancer (EXACT). Pilot Feasibility Stud. 2019 Aug 16;5:102. doi: 10.1186/s40814-019-0486-6. eCollection 2019. PMID 31428443